CLINICAL TRIAL: NCT03879850
Title: Perioperative Electroencephalography Characteristics of Postoperative Delirium in Elderly
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsche Forschung (Projekt No 409495393) (Unknown)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: EPOD
Record Dates: First submitted 2019-02-25; First posted 2019-03-19 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propofol group: This is a prospective, observational study in surgical patients undergoing elective surgery under general anesthesia stratified for the anesthetic agent used intraoperatively - i.v. Propofol - focusing on pre-, intra- and postoperative EEG spectral parameters in elderly patients.
- Volatile group: This is a prospective, observational study in surgical patients undergoing elective surgery under general anesthesia stratified for the anesthetic agent used intraoperatively - volatile anesthetic agent as Sevoflurane or Desflurane - focusing on pre-, intra- and postoperative EEG spectral parameters in elderly patients.

SUMMARY:
The investigators aim to identify preoperative Electroencephalogram (EEG) markers indicating patients at risk to develop postoperative delirium (POD), so that the anesthetist may adjust medications and dosages in order to avoid POD. Second, the investigators aim to specify intraoperative EEG signatures and EEG states that are related to POD and long-term cognitive dysfunction, again to enable physicians to adapt their procedure. Third, the investigators aim to identify EEG signatures during stay in the recovery room that is directly related to POD, and may therefore be used as diagnostic tool, as well as a predictor for the development of long-term cognitive deficits (POCD).

DETAILED DESCRIPTION:
The investigators conduct this observational study to identify pre-, intra- and postoperative Electroencephalogram (EEG) signatures / intraoperative EEG states related to postoperative delirium (POD) and postoperative cognitive deficit (POCD) in elderly patients > 70 years. This includes the following tasks at five different time-points

1. Pre-operative frontal EEG recording during anesthesia evaluation one day before surgery / anesthesia to develop an EEG marker to predict the development of POD. This includes the stratification of EEG data related to age, gender, and pre-operative cognitive function. Pre-operative POCD assessment (CANTAB connect, word pair recognition test, Mini Mental State Test, and Trail Making Test A and B) to classify cognitive capacity of each patient before start of anesthesia.
2. Intra-operative frontal EEG recording from start of anesthesia procedure until discharge to the recovery room to identify EEG signatures / EEG states to predict the development of POD / POCD. This includes the stratification of EEG data related to age, gender, pre-medication, anesthetics, and analgesics used during anesthesia procedure.
3. Post-operative frontal EEG recording during the recovery room stay to develop an EEG marker / identify EEG signatures to diagnose POD and predict POCD. This includes the stratification of EEG data related to age, gender, anesthesia procedure, and analgesics administered during the recovery room stay. POD will be assessed during stay in the recovery room by the NuDesc Score and DSM V criteria.
4. Follow-up POD assessments until the 5th postoperative day, where the patient will be visited twice daily (8a.m.-10a.m. and 5p.m.-7p.m.) and assessed via DSM V / NuDesc criteria on the peripheral ward, or via Confusion Assessment Method for intensive Care Unit (CAM-ICU) criteria during an intensive care unit stay.
5. Follow-up POCD assessments one day before and 3 months after surgery, where the patient will undergo a ~1 hour cognitive testing with the CANTAB connect.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >70 years
* Planned operation time >1 hour
* Expected hospital treatment period of 5 days,
* Anesthesia induction, anesthesia maintenance with either Propofol or an inhalative anesthetic agent as Sevoflurane or Desflurane,
* The ability to give informed consent

Exclusion Criteria:

* Patients with a history of neurological or psychiatric disorders
* Known carotid artery Stenosis
* Obstructive sleep apnea Syndrome
* Planned neurosurgery
* Current medication of tranquilizers / antidepressants
* Isolation of patients with multi-resistant Bacteria
* Inability of the patients to speak and/or read German
* Homelessness or other circumstances where the patient would not be reachable by phone or postal services during follow-up
* Intraoperative EEG data file analysis will be excluded ex post,

  1. when intraoperative use of any other anesthetic agent for induction as Propofol occurred or
  2. by use of any other anesthetic agent for anesthesia maintenance other than Propofol or volatile anesthetics as Sevoflurane or Desflurane or
  3. when anesthesia agents as Ketamine, Nitrous oxide, Etomidate or Dexmedetomidine were given or
  4. if body temperature drops below 34° or rises above 38° during surgery

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This is a prospective, observational study in surgical patients undergoing elective surgery under general anesthesia stratified for the anesthetic agent used intraoperatively - i.v. Propofol (Propofol group) or volatile anesthetic agent as Sevoflurane or Desflurane (Volatile group) - focusing on pre-, intra- and postoperative EEG spectral parameters in elderly patients.
Sampling Method: Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Delirium- Diagnostic and Statistical Manual of Mental Disorders (DSM-V) | Patients will be follow until hospital discharge, or maximal until postoperative day 5
  Postoperative delirium rate, defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
Incidence of Postoperative Delirium - Nursing Delrium Scale (Nu-DESC) | Patients will be follow until hospital discharge, or maximal until postoperative day 5
  Postoperative delirium rate, defined according to ≥ 2 cumulative points in the nursing Delirium Screening Scale (Nu-DESC)
Incidence of Postoperative Delirium - Intensive Care Unit (CAM-ICU) | Patients will be followed on intensive care unit until hospital discharge, or maximal until postoperative day 5
  Postoperative delirium rate, defined according to positive Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score
Incidence of Postoperative Delirium - Confusion Assessment Method (CAM) | Patients will be followed on peripheral ward until hospital discharge, or maximal until postoperative day 5
  Postoperative delirium rate, defined according to positive Confusion Assessment Method (CAM)

SECONDARY OUTCOMES:
Incidence of postoperative cognitive deficit (POCD) - CANTAB | Up to 3 months
  POCD will be measured by a defined Cambridge Neuropsychological Test Automated Battery (CANTAB) on the day before the operation and after 3 months
Incidence of postoperative cognitive deficit (POCD) - MMSE | Up to 3 months
  POCD will be measured by Mini Mental State Examination (MMSE) on the day before the Operation, on day 5 and after 3 months
Incidence of Neurocognitive disorder | Up to 3 months
  Neurocognitive Disorder is evaluated according to DSM-V (postoperative cognitive deficit, activities of daily living, instrumental activities of daily living, subjective memory sensing.
Incidence of postoperative cognitive deficit (POCD) - Word pair recognition test | Up to 5 days
  POCD will be measured by Nürnberger-Altersinventar-Test - word pair recognition test on the day before the operation, day 1 ,3 and 5
Post-operative, bi-frontal alpha-band power | Up to discharge from the recovery room
  Bi-frontal EEG recording with surface electrodes (Fp1, Fp2, F7 and F8), Spectral analysis by Matlab code
Bi-frontal overall EEG band power | Up to discharge from the recovery room
  Postoperative bi-frontal EEG recording with surface electrodes (Fp1, Fp2, F7 and F8), Spectral analysis by Matlab code
Burst suppression duration | During anesthesia procedure
  Intraoperative bi-frontal EEG recording with surface electrodes (Fp1, Fp2, F7 and F8), raw EEG analysis
Pain monitoring | During anesthesia procedure
  Intraoperative pain monitoring is measured by Nociception Level Index (NOL
Duration of Delirium (DSM-V) | Participants will be followed for the duration of hospital stay, or maximal until postoperative day 5
  Postoperative duration of delirium, defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
Duration of Delirium (Nu-DESC) | Participants will be followed for the duration of hospital stay, or maximal until postoperative day 5
  Postoperative duration of delirium, defined according to Nursing Delirium Screening Scale (Nu-DESC)
Duration of Delirium (CAM-ICU) | Participants will be followed for the duration of hospital stay, or maximal until postoperative day 5
  Postoperative duration of delirium, defined according to Confusion Assessment Method for the Intensive Care Unit (CAM-ICU)Confusion Assessment Method (CAM), Chart Review
Duration of Delirium (CAM) | Participants will be followed for the duration of hospital stay, or maximal until postoperative day 5
  Postoperative duration of delirium, defined according to Confusion Assessment Method (CAM)
Intensive care unit length of stay | Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
  Intensive care unit length of staywill be assessed by chart review at hospital discharge.
Hospital length of stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Hospital length of stay will be assessed by chart review at 3 months.
Mortality | Up to 3 months
  Mortality will be assessed by chart review at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No